CLINICAL TRIAL: NCT00745875
Title: A Phase II, Double-blind, Placebo Controlled, Randomised Study to Assess the Efficacy and Safety of ZD4054 (Zibotentan) in Combination With Pemetrexed (Alimta®) vs. Pemetrexed Alone in Patients With Non-small Cell Lung Cancer Who Have Failed One Prior Platinum-based Chemotherapy Regimen
Brief Title: ZD4054 (Zibotentan) Phase II Non-Small Cell Lung Cancer Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D4320C00035
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2012-06-06 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-04

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
Keywords: NSCLC; Phase II; ZD4054; Pemetrexed; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — ZD4054; Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): ZD4054 + Pemetrexed
  Interventions: Drug: ZD4054; Drug: Pemetrexed
- 2 (Placebo Comparator): ZD4054 matched placebo + pemetrexed
  Interventions: Drug: Pemetrexed; Drug: Placebo

INTERVENTIONS:
Drug: ZD4054 — 10mg oral tablet, once daily
  Other Names: Zibotentan
  Arms: 1
Drug: Pemetrexed — 500mg2/m IV infusion
  Other Names: Alimta
Drug: Placebo — 10mg oral tablet, once daily
  Arms: 2

SUMMARY:
The aim of this study is to collect initial efficacy and safety data on the use of a new treatment ZD4054 (Zibotentan) when used in combination with pemetrexed (a standard chemotherapy agent) for the treatment of non-small cell lung cancer compared to treatment with pemetrexed alone

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic NSCLC on entry into study suitable for pemetrexed therapy
* Patients that meet one of the following criteria: - progressed following one prior platinum-based chemotherapy regimen for locally advanced or metastatic disease; -progressed within 6 months of adjuvant platinum-based chemotherapy
* Life expectancy of > 12 weeks

Exclusion Criteria:

* Prior treatment with pemetrexed in the last 12 months.
* Prior therapy with an ET receptor antagonist
* Any recent surgery, unhealed surgical incision, severe concomitant medical condition (eg, unstable cardiac, hepatic or renal disease) or significant laboratory finding which makes it undesirable for the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-08; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Morris, MD, Study Director — AstraZeneca; Christos Chouaid, MD, Prof, Principal Investigator — Hospital Saint-Antoine, Cedex, France
Locations (13):
- Bulgaria (3):
  - research Site, Pleven
  - Research Site, Sofia
  - Research Site, Varna
- Czechia (2):
  - Research Site, Jičín
  - Research Site, Prague
- France (2):
  - Research Site, Cedex
  - Research Site, Strasbourg
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
- Ukraine (4):
  - Research Site, Chernivtsi
  - Research Site, Kiev
  - Research Site, Sumy
  - Research Site, Uzngorod

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 patients with locally advanced or metastatic non-small cell lung cancer (NSCLC) where the histology was not predominantly of squamous type were recruited between 12th August 2008 and 3rd June 2009.
Pre-assignment Details: 14 of the 80 enrolled patients were not randomised to treatments groups: 7 patients did not meet one or more of the study inclusion or exclusion criteria, 3 patients failed screening, 2 patients were not included due to investigator decision, 1 patient withdrew consent and 1 patient died.
Groups:
- Placebo + Pemetrexed: Pemetrexed 500 mg/m2 Intravenous (IV) infusion every 21 days + placebo oral tablet once daily
- ZD4054 + Pemetrexed: ZD4054 10 mg oral tablet once daily + Pemetrexed 500 mg/m2 IV infusion every 21 days
Period: Overall Study
Arm/Group | Placebo + Pemetrexed | ZD4054 + Pemetrexed
Started | 36 (Started - Number of patients randomised) | 30 (Started - Number of patients randomised)
Completed | 32 (Completed - Number of patients discontinued study treatment at data cut-off (17th January 2010)) | 26 (Completed - Number of patients discontinued study treatment at data cut-off (17th January 2010))
Not Completed | 4 | 4
Not completed — Continuing study treatment | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo + Pemetrexed | ZD4054 + Pemetrexed | Total
Number analyzed (Participants) | 36 | 30 | 66
Age Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (12.06) | 57.5 (10.44) | 57 (11.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 28 | 19 | 47

OUTCOME MEASURES:

1. Primary Outcome: Time to Death
Description: Median time (in days) from randomisation until death using the Kaplan-Meier method (Calculator for survival probability)
Time Frame: Patients were followed up for survival every week for the first 3 weeks then every 3 weeks whilst on study medication until the data cut-off (17th January 2010).
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo + Pemetrexed | ZD4054 + Pemetrexed
Number analyzed (Participants) | 36 | 30
Days | 193 [27 to 437] | 146 [19 to 427]

2. Secondary Outcome: Progression-free Survival
Description: Median time (in days) from randomisation until disease progression/death using the Kaplan-Meier method
Time Frame: Tumour assessments for progression were performed at screening, every 3 weeks, Mandatory Tumour Assessment Visit (19 August 2009 ± 3 days), treatment discontinuation
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo + Pemetrexed | ZD4054 + Pemetrexed
Number analyzed (Participants) | 36 | 30
Days | 87 [27 to 283] | 110 [18 to 303]

ADVERSE EVENTS:
Arm/Group | Placebo + Pemetrexed | ZD4054 + Pemetrexed
Serious Adverse Events (participants affected / at risk) | 7/30 | 4/36
Other Adverse Events (participants affected / at risk) | 22/30 | 20/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Pemetrexed (N=30) | ZD4054 + Pemetrexed (N=36)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Right Ventricular Failure (Cardiac disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Adverse Drug Reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 0 | 1
Metastases To Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Pemetrexed (N=30) | ZD4054 + Pemetrexed (N=36)
Anaemia (Blood and lymphatic system disorders) | 8 | 7
Neutropenia (Blood and lymphatic system disorders) | 5 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Oedema Peripheral (General disorders) | 1 | 4
Fatigue (General disorders) | 1 | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 0
Bacterial Infection (Infections and infestations) | 2 | 0
Body Temperature Increased (Infections and infestations) | 3 | 2
Brain Natriuretic Peptide Increased (Infections and infestations) | 0 | 3
Weight Decreased (Infections and infestations) | 3 | 3
Alanine Aminotransferase Increased (Infections and infestations) | 2 | 2
Aspartate Aminotransferase Increased (Infections and infestations) | 1 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AstraZeneca can review results communications prior to public release and may within 60 days of receipt require amendments to be made. AstraZeneca can also require that submission or disclosure be delayed for 90 days to allow for the filing of a patent application.